CLINICAL TRIAL: NCT06858319
Title: A Multicenter Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of Zigakibart in Adults With Primary IgA Nephropathy.
Brief Title: Open-label Extension Study of Zigakibart in Adults With IgA Nephropathy.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFUB523A12302B
Record Dates: First submitted 2025-02-21; First posted 2025-03-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Kidney Diseases; Kidney Diseases, Chronic; Urological Diseases; Glomerulonephritis; Glomerular Disease; Glomerulonephritis, IGA; Glomerulopathy; Immunoglobulin Disease
Keywords: Urologic Diseases; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Male Urogenital Diseases; Glomerulonephritis; Nephritis; Autoimmune Diseases; Immune System Diseases; Kidney Diseases; Glomerulonephritis, IGA; Primary IgA / Immunoglobulin A nephropathy; eGFR; UPCR; UACR; FUB523
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Urologic Diseases; Glomerulonephritis; Glomerulonephritis, IGA; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Male Urogenital Diseases; Nephritis; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- zigakibart (Experimental): Participants will receive zigakibart.
  Interventions: Drug: zigakibart

INTERVENTIONS:
Drug: zigakibart — solution for subcutaneous injection
  Other Names: FUB523; BION-1301

SUMMARY:
The purpose of this study is to determine if zigakibart is safe and effective for long-term use in patients with immunoglobulin A nephropathy (IgAN). This is an extension study for patients who have already completed an another zigakibart study.

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, open-label extension (OLE) study to Phase 3, randomized CHK02-02 (CFUB523A12301)-BEYOND clinical study, Phase 1/2 ADU-CL-19 (CFUB523A12103) clinical study, and any other Novartis-sponsored clinical study of zigakibart in IgAN.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the OLE study.
2. Completion of the parent study (both participants assigned to receive the investigational product and placebo) as defined by the respective protocol.
3. Per Investigator's clinical judgment, the participant may benefit from receiving open-label treatment of zigakibart 600 mg s.c. Q2W.

Exclusion Criteria:

1. Participants who prematurely withdrew from zigakibart parent studies in IgAN for any reason.
2. Participants who at the time of first study treatment administration in the OLE are receiving chronic dialysis (≥30 days) or who require kidney transplantation.
3. Acute kidney injury (AKI), defined by AKIN criteria (Mehta et al 2007) within 4 weeks of first study treatment administration in the OLE study.
4. Clinical suspicion or diagnosis of rapidly progressive glomerulonephritis (RPGN), defined by KDIGO guidelines, or another glomerulopathy at the time of first study treatment administration in the OLE study.
5. Received a live vaccination within 12 weeks prior to first study treatment administration in the OLE study or plan to have a live vaccination within 6 months after the last dose of study treatment.
6. Use of systemic corticosteroid therapy (including budesonide) or other immunosuppressive therapy such as but not limited to mycophenolate, azathioprine, cyclosporine, tacrolimus, cyclophosphamide, etc., and herbs such as Tripterygium Wilfordii Hook F, Caulis sinomenii, and Sinomenium acutum for > 2 weeks in the 12 weeks prior to first study treatment administration in the OLE study; use of rituximab within 180-days of first study treatment administration in the OLE study.
7. Current severe infection at the time of first study treatment in the OLE study or history of recurrent, severe, infections as determined by the Investigator.
8. Newly diagnosed positive serology for hepatitis A virus IgM antibodies (anti-HAV IgM), hepatitis B surface antigen (HBsAg), detectable hepatitis B virus (HBV) DNA, hepatitis C virus (HCV) antibodies (participants who completed treatment and are persistently antibody positive but have documentation of negative HCV polymerase chain reaction [PCR] will be allowed), or antibodies to HIV-1 and/or HIV-2.
9. Newly diagnosed malignancy (participants with basal cell carcinoma that was completely resected or curatively treated cervical carcinoma in situ or low-risk prostate cancer (i.e., Gleason score < 7 and prostate specific antigen < 10 ng/mL) are eligible for the study).
10. Pregnancy or breastfeeding or intent to become pregnant or to donate sperm during the study period and until 24 weeks after last dose.
11. History or evidence of any other clinically significant medical or psychiatric disorder, condition, disease, or laboratory finding that, in the discretion of the Investigator, constitutes an uncertain or unfavorable benefit-risk for continued long-term therapy with zigakibart.
12. Confirmed IgG levels < 3 g/L prior to first study treatment administration in the OLE study.
13. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, from menarche until becoming post-menopausal unless they are using highly effective methods of contraception (failure rate < 1% per year) while taking study treatment and for 24 weeks after stopping study treatment. Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., hormonal profile confirming menopause and/or age-appropriate history of vasomotor symptoms).
14. Sexually active males unwilling to use a highly effective methods of contraception during intercourse while taking study treatment and for 24 weeks after stopping study treatment. In addition, male participants must not donate sperm for the time period specified above.

Highly effective contraception methods for both women and men include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Note that periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Bilateral oophorectomy with or without hysterectomy, total hysterectomy or bilateral salpingectomy at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment are they considered to be not of childbearing potential.
* Bilateral tubal occlusion, bilateral tubal ligation (at least six weeks before taking study treatment).
* Sterilization (vasectomy) of male partner(s) of the female participant at least 6 months prior to first study treatment provided partner(s) has(have) received medical confirmation of surgical success.
* Use of hormonal contraception methods:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation; oral, intravaginal or transdermal.
* Progestogen-only hormonal contraception (where inhibition of ovulation is not the primary or only mode of action): oral, injectable or implantable.
* Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS). In case of use of hormonal contraception, women should have been stable on the same method for a minimum of 3 months before taking study treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2031-06-25 (Estimated); Study Completion 2031-06-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events. | Date of first administration of study treatment to 24 weeks after the date of the last actual administration of study treatment
  Number of participants with adverse events will be provided.
Number of participants with serious adverse events. | Date of first administration of study treatment to 24 weeks after the date of the last actual administration of study treatment
  Number of participants with serious adverse events will be provided.
Number of participants with adverse events of special interest. | Date of first administration of study treatment to 24 weeks after the date of the last actual administration of study treatment
  Number of participants with adverse events of special interest will be provided.

SECONDARY OUTCOMES:
Change in UPCR from Baseline to Week 48 and Week 96. | Baseline visit, Week 48 and Week 96.
  The change in the ratio of urine protein to urine creatinine (UPCR), based on 24-hour urine collection, from Baseline to Week 48 and to Week 96.
Change in eGFR from Baseline to Week 96. | Baseline visit and Week 96.
  Estimated glomerular filtration rate (eGFR) will be calculated using the chronic kidney disease-epidemiology collaboration (CKD-EPI) creatinine equation. The change (difference) in eGFR between Baseline and Week 96 timepoints will then be calculated.
Change in eGFR from BEYOND parent study Baseline to Week 96 of OLE study. | Baseline visit and Week 96.
  eGFR will be calculated using the chronic kidney disease-epidemiology collaboration (CKD-EPI) creatinine equation. The change (difference) in eGFR between Baseline in the BEYOND study and Week 96 in OLE study will then be calculated.
Serum concentration values of zigakibart at scheduled visits. | Baseline visit, Week 24 and Week 96.
  Serum concentration values will be provided for the following scheduled visits: Day 1, Week 24 and Week 96.
Change from baseline in Immunoglobulin (IgA, IgG and IgM) levels. | Baseline visit, Week 2, Week 4, Week 24, Week 48, Week 72, Week 96, then every 24 weeks after Week 96 through EOT.
  Immunoglobulin (IgA, IgG and IgM) levels will be assessed from samples collected at Week 2, Week 4, Week 24, Week 48, Week 72, Week 96, then every 24 weeks after Week 96 through EOT. The change (difference) in immunoglobulin levels between Baseline and the noted timepoints will then be calculated.
Presence of circulating binding and neutralizing anti- drug antibodies (ADA/Nab). | Baseline visit, Week 24 and Week 96.
  Number of participants with circulating binding and neutralizing anti-drug antibodies (ADA/Nab) in blood will be provided at the following scheduled visits: Day 1, Week 24, Week 96.
Number of participants with abnormal safety laboratory parameters. | Date of first administration of study treatment to the date that study treatment is discontinued, assessed up to approximately 5 years.
  Number of participants with abnormal safety laboratory parameters will be provided.
Number of participants with abnormal vital sign measurements. | Date of first administration of study treatment to the date that study treatment is discontinued, assessed up to approximately 5 years.
  Number of participants with abnormal vital sign measurements will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (3):
  - Colorado Kidney Care Nephrology, Denver, Colorado
  - NY Nephrology, Clifton Park, New York
  - Knoxville Kidney Center Pllc, Brentwood, Tennessee
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Santa Fe
- Novartis Investigative Site, Seoul, Korea, South Korea